CLINICAL TRIAL: NCT00670540
Title: A Prospective Epidemiological Multicenter Cohort Study on Patients Clinically Suspected of Deep Vein Thrombosis or Pulmonary Embolism
Brief Title: Epidemiology of Thromboembolism Disease: A Cohort Study
Acronym: OPTIMEV
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Sanofi (Industry); Ministry of Health, France (Other Government); SFMV (Société Française de Médecine Vasculaire) (Unknown)
Responsible Party: Sponsor
Other Study IDs: DCIC-04-02
Record Dates: First submitted 2008-04-30; First posted 2008-05-02 (Estimated); Results first posted 2012-05-03 (Estimated); Last update posted 2012-05-08 (Estimated); Status verified 2012-05

CONDITIONS: Vascular Diseases; Embolism and Thrombosis; Phlebitis; Venous Insufficiency; Pulmonary Embolism
Keywords: pulmonary embolism; duplex ultrasound examination; recurrence
MeSH Terms: conditions — Vascular Diseases; Embolism and Thrombosis; Phlebitis; Venous Insufficiency; Pulmonary Embolism; Recurrence | interventions — vinyltriethoxysilane

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: patients with suspected Deep Vein Thrombosis (DVT) or Pulmonary Embolism (PE)
  Interventions: Other: procedure of Deep Vein Thrombosis (DVT) and PE (Pulmonary Embolism) diagnosis

INTERVENTIONS:
Other: procedure of Deep Vein Thrombosis (DVT) and PE (Pulmonary Embolism) diagnosis — patients with a clinical suspicion of Venous ThromboEmbolism (VTE = Deep Vein Thrombosis or Pulmonary Embolism) were eligible
  Other Names: VTE (venous thromboembolism); DVT (deep vein thrombosis); PE (pulmonary embolism)

SUMMARY:
The purpose of this study is to determine different risk factors of thromboembolic disease. Different points will be studied

1. do different types of thromboembolic disease (distal Deep Vein Thrombosis (DVT), proximal DVT, Pulmonary Embolism (PE) and DVT, PE without DVT) have the same clinical significance (risk factors and prognosis) ?
2. Is it necessary to obtain a detailed history of thromboembolic disease ?
3. Do older patients have particular risk factors ?
4. Do preventive treatments modify the level of risk factors and the clinical signs of thromboembolic disease ?
5. Do predictive clinical scores have the same performance for both in and outpatients ?
6. Can patients with a potential high level of thromboembolic risk (surgery, pregnancy) but no clinical thromboembolic symptoms, develop a low risk ?
7. The evolution of the disease in patients with negative or positive Venous ThromboEmbolism (VTE) exploratory tests.

DETAILED DESCRIPTION:
The OPTIMEV study is a prospective epidemiological multicenter cohort study, including in-and outpatients clinically suspected of thromboembolic disease. Deep vein thrombosis is diagnosed using a duplex ultrasound examination, whereas pulmonary embolism is investigated by lung scan scintigraphy or computed helical tomodensitometry and/or duplex ultrasound examination. Initial data on medical history, clinical symptoms, presence of transient and chronic risk factors, diagnosis at the end of the medical examination, diagnostic tests results, treatment (type and duration) are collected by the physician into an electronic medical record. Other general medical considerations are collected (particularly on cardiovascular diseases). A phone follow up at 3 months, 1, 2 and 3 years is realised by the Centre for Clinical Research of Grenoble. All Venous ThromboEmbolism (VTE) positive patients (including superficial vein thrombosis) are contacted. For each VTE positive a negative one is selected (same site, same season). Data on mortality, development or recurrence of VTE, treatments prescribed (type + duration), major bleeding, cancer onset, cardiovascular events and venous insufficiency (leg ulcer) are collected. All these serious adverse events are documented and reviewed by an independent critical events committee.

ELIGIBILITY:
Inclusion Criteria:

* patient aged more than 18
* male or female
* patients with clinical thromboembolic signs (deep vein thrombosis or pulmonary embolism)

Exclusion Criteria:

* patient less than 18 years old
* patient unable to understand
* patient who refused to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All male or female inpatients and outpatients hospital and office-based. 18 years old with clinical suspicion of deep vein thrombosis (DVT) or pulmonary embolism (PE).
  Patients with cognitive disorders or language impairment preventing collection of risk factor data by history-taking were excluded.
Sampling Method: Non-Probability Sample
Enrollment: 8256 (Actual)
Dates: Start 2004-11; Primary Completion 2009-01 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean Luc JB BOSSON, MD, Principal Investigator — University Hospital, Grenoble; Marie Antoinette SEVESTRE, MD, Study Chair — Amiens University Hospital
Locations (231):
- University Hospital ND des Bruyeres Liege, Chênée, Belgium
- France (229):
  - General Hospital, Abbeville
  - Office-based Specialist in vascular medecine, Albertville
  - Office-based Specialist in vascular medecine, Albi
  - Office-based Specialist in vascular medecine, Alençon
  - Office-based Specialist in vascular medecine, Alès
  - Office-based Specialist in vascular medecine, Ambares
  - Office-based Specialist in vascular medecine, Amberieu En Buget
  - Office-based Specialist in vascular medecine, Amiens
  - University Hospital, Amiens
  - Office-based Specialist in vascular medecine, Ancenis
  - Office-based Specialist in vascular medecine, Angers
  - University Hospital, Angers
  - Office-based Specialist in vascular medecine, Annecy
  - Hospital, Annecy
  - Hospital, Armentières
  - Office-based Specialist in vascular medecine, Arnouville
  - Office-based Specialist in vascular medecine, Arpajon
  - Office-based Specialist in vascular medecine, Arras
  - Office-based Specialist in vascular medecine, Aubenas
  - Hospital, Auch
  - Office-based Specialist in vascular medecine, Auxerre
  - Office-based Specialist in vascular medecine, Bagnoles-de-l'orme
  - Office-based Specialist in vascular medecine, Beauvais
  - University Hospital, Belfort
  - Office-based Specialist in vascular medecine, Bergerac
  - Office-based Specialist in vascular medecine, Besançon
  - Office-based Specialist in vascular medecine, Béziers
  - Office-based Specialist in vascular medecine, Blagnac
  - Office-based Specialist in vascular medecine, Bordeaux
  - Hospital St ANDRE, Bordeaux
  - Office-based Specialist in vascular medecine, Boulogne-sur-Mer
  - Office-based Specialist in vascular medecine, Bourg-en-Bresse
  - Office-based Specialist in vascular medecine, Bourgoin
  - Office-based Specialist in vascular medecine, Brest
  - University Hospital La Cavale Blanche, Brest
  - Office-based Specialist in vascular medecine, Bretenoux
  - Office-based Specialist in vascular medecine, Brétigny-sur-Orge
  - Office-based Specialist in vascular medecine, Bron
  - Office-based Specialist in vascular medecine, Cabestany
  - University Hospital, Caen
  - Office-based Specialist in vascular medecine, Caluire-et-Cuire
  - Office-based Specialist in vascular medecine, Cambrai
  - Office-based Specialist in vascular medecine, Cannes
  - Office-based Specialist in vascular medecine, Carcassonne
  - Hospital Antoine Gayraud, Carcassonne
  - Office-based Specialist in vascular medecine, Castanet-Tolosan
  - Office-based Specialist in vascular medecine, Castres
  - Office-based Specialist in vascular medecine, Cenon
  - Office-based Specialist in vascular medecine, Chalon En Champagne
  - Office-based Specialist in vascular medecine, Chalon-sur-Saône
  - Office-based Specialist in vascular medecine, Chambéry
  - Hospital, Chambéry
  - Office-based Specialist in vascular medecine, Champagnole
  - Office-based Specialist in vascular medecine, Chantilly
  - Office-based Specialist in vascular medecine, Charleville-Mézières
  - Office-based Specialist in vascular medecine, Chartres
  - Office-based Specialist in vascular medecine, Châteaubriant
  - Office-based Specialist in vascular medecine, Cholet
  - Office-based Specialist in vascular medecine, Clamart
  - Office-based Specialist in vascular medecine, Clapiers
  - Office-based Specialist in vascular medecine, Clermont-Ferrand
  - Hospital Hotel Dieu, Clermont-Ferrand
  - Office-based Specialist in vascular medecine, Clermont-l'Hérault
  - Office-based Specialist in vascular medecine, Clisson
  - Office-based Specialist in vascular medecine, Cluses
  - Office-based Specialist in vascular medecine, Colomiers
  - General Hospital, Compiègne
  - Office-based Specialist in vascular medecine, Coulommiers
  - Office-based Specialist in vascular medecine, Crolles
  - Office-based Specialist in vascular medecine, Denain
  - Office-based Specialist in vascular medecine, Dieppe
  - Office-based Specialist in vascular medecine, Dijon
  - Hospital Bocage, Dijon
  - University Hospital, Dijon
  - Office-based Specialist in vascular medecine, Draguignan
  - Office-based Specialist in vascular medecine, Ermont
  - Office-based Specialist in vascular medecine, Échirolles
  - Office-based Specialist in vascular medecine, Évreux
  - Office-based Specialist in vascular medecine, Feytiat
  - Office-based Specialist in vascular medecine, Fécamp
  - Office-based Specialist in vascular medecine, Figeac
  - Hospital, Flers
  - Office-based Specialist in vascular medecine, Foix
  - Hospital Val d'Ariege, Foix
  - Office-based Specialist in vascular medecine, Fontenay-le-Comte
  - Office-based Specialist in vascular medecine, Glanes
  - Office-based Specialist in vascular medecine, Grenoble
  - University Hospital Grenoble, Grenoble
  - Office-based Specialist in vascular medecine, Gruchet-le-Valasse
  - Office-based Specialist in vascular medecine, Hœnheim
  - Office-based Specialist in vascular medecine, Issy-les-Moulineaux
  - Office-based Specialist in vascular medecine, Istres
  - Office-based Specialist in vascular medecine, L'Île-Rousse
  - Office-based Specialist in vascular medecine, La Roche-sur-Yon
  - Departemental Hospital, La Roche-sur-Yon
  - Office-based Specialist in vascular medecine, La Rochelle
  - Office-based Specialist in vascular medecine, Lannion
  - Office-based Specialist in vascular medecine, Lattes
  - Office-based Specialist in vascular medecine, Laval
  - Office-based Specialist in vascular medecine, Laxou
  - Hospital Versailles, Le Chesnay
  - Office-based Specialist in vascular medecine, Le Mans
  - Office-based Specialist in vascular medecine, Le Quesnoy
  - Office-based Specialist in vascular medecine, Levallois-Perret
  - Office-based Specialist in vascular medecine, Limoges
  - Office-based Specialist in vascular medecine, Lisieux
  - Hospital Saint Philibert, Lomme
  - Office-based Specialist in vascular medecine, Longjumeau
  - Office-based Specialist in vascular medecine, Longwy
  - Office-based Specialist in vascular medecine, Lons-le-Saunier
  - Office-based Specialist in vascular medecine, Lorient
  - Office-based Specialist in vascular medecine, Louviers
  - Hospital Edouard Herriot, Lyon
  - University Hospital, Lyon
  - Office-based Specialist in vascular medecine, Malemort-sur-Corrèze
  - Office-based Specialist in vascular medecine, Manosque
  - Office-based Specialist in vascular medecine, Mantes-la-Jolie
  - Office-based Specialist in vascular medecine, Marcq-en-Barœul
  - Office-based Specialist in vascular medecine, Marseille
  - Office-based Specialist in vascular medecine, Martinique
  - Office-based Specialist in vascular medecine, Maurepas
  - Office-based Specialist in vascular medecine, Meaux
  - Office-based Specialist in vascular medecine, Metz
  - Office-based Specialist in vascular medecine, Meudon
  - Office-based Specialist in vascular medecine, Moissac
  - Office-based Specialist in vascular medecine, Montaigu
  - Office-based Specialist in vascular medecine, Montbéliard
  - General Hospital, Montbéliard
  - Hospital Jacques Monod, Montivilliers
  - Office-based Specialist in vascular medecine, Montluçon
  - Hospital, Montluçon
  - Hospital, Montmorillon
  - Office-based Specialist in vascular medecine, Montpellier
  - Hospital St Eloi, Montpellier
  - Office-based Specialist in vascular medecine, Mulhouse
  - Office-based Specialist in vascular medecine, Nancy
  - Office-based Specialist in vascular medecine, Nantes
  - Office-based Specialist in vascular medecine, Narbonne
  - Office-based Specialist in vascular medecine, Nice
  - Office-based Specialist in vascular medecine, Niort
  - Office-based Specialist in vascular medecine, Nîmes
  - Office-based Specialist in vascular medecine, Noumea (Nouvelle Calédonie)
  - Office-based Specialist in vascular medecine, Noyal-Pontivy
  - Office-based Specialist in vascular medecine, Noyon
  - Office-based Specialist in vascular medecine, Orange
  - Regional Hospital, Orleans La Source
  - Office-based Specialist in vascular medecine, Orléans
  - Office-based Specialist in vascular medecine, Paris
  - Hospital Croix Saint Simon, Paris
  - Office-based Specialist in vascular medecine, Pessac
  - Hospital, Périgueux
  - Office-based Specialist in vascular medecine, Péronne
  - Office-based Specialist in vascular medecine, Poissy
  - Office-based Specialist in vascular medecine, Poitiers
  - Office-based Specialist in vascular medecine, Pontarlier
  - Office-based Specialist in vascular medecine, Pornic
  - Office-based Specialist in vascular medecine, Puilboreau
  - Office-based Specialist in vascular medecine, Quimper
  - Office-based Specialist in vascular medecine, Rambouillet
  - Office-based Specialist in vascular medecine, Redon
  - Office-based Specialist in vascular medecine, Reims
  - University Hospital, Reims
  - Office-based Specialist in vascular medecine, Riom
  - Office-based Specialist in vascular medecine, Rivesaltes
  - Office-based Specialist in vascular medecine, Rochefort
  - Office-based Specialist in vascular medecine, Rodez
  - Hospital, Rodez
  - Office-based Specialist in vascular medecine, Romans-sur-Isère
  - Office-based Specialist in vascular medecine, Rouen
  - Office-based Specialist in vascular medecine, Sablé-sur-Sarthe
  - Office-based Specialist in vascular medecine, Saint Genevieve Des Bois
  - Cmc Les Petites Roches, Saint Hilaire Du Touvert
  - Office-based Specialist in vascular medecine, Saint Pierre (ile de La Reunion)
  - Office-based Specialist in vascular medecine, Saint-Aubin-de-Médoc
  - Office-based Specialist in vascular medecine, Saint-Benoît
  - Office-based Specialist in vascular medecine, Saint-Brieuc
  - Office-based Specialist in vascular medecine, Saint-Chamond
  - Office-based Specialist in vascular medecine, Saint-Cloud
  - Office-based Specialist in vascular medecine, Saint-Cyr-l'École
  - Office-based Specialist in vascular medecine, Saint-Etienne
  - University Hospital, Saint-Etienne
  - Office-based Specialist in vascular medecine, Saint-Égrève
  - Office-based Specialist in vascular medecine, Saint-Gaudens
  - Office-based Specialist in vascular medecine, Saint-Germain-en-Laye
  - Office-based Specialist in vascular medecine, Saint-Lô
  - Memorial Hospital, Saint-Lô
  - Office-based Specialist in vascular medecine, Saint-Martin-Boulogne
  - Office-based Specialist in vascular medecine, Saint-Priest
  - Hospital, Saint-Quentin
  - Office-based Specialist in vascular medecine, Sallanches
  - Office-based Specialist in vascular medecine, Salon-de-Provence
  - Office-based Specialist in vascular medecine, Sarcelles
  - Office-based Specialist in vascular medecine, Sarrebourg
  - Office-based Specialist in vascular medecine, Sarreguemines
  - Office-based Specialist in vascular medecine, Saverne
  - Office-based Specialist in vascular medecine, Savigny-sur-Orge
  - Office-based Specialist in vascular medecine, Sceaux
  - Office-based Specialist in vascular medecine, Sèvres
  - Office-based Specialist in vascular medecine, Sélestat
  - Office-based Specialist in vascular medecine, Strasbourg
  - Regional University Hospital, Strasbourg
  - Office-based Specialist in vascular medecine, Talant
  - Office-based Specialist in vascular medecine, Tarare
  - Office-based Specialist in vascular medecine, Toulouse
  - University Hospital Rangueil Larrey, Toulouse
  - University Hospital Rangueil, Toulouse
  - University Hospital, Toulouse
  - Office-based Specialist in vascular medecine, Tours
  - Office-based Specialist in vascular medecine, Trois Rivieres (guadeloupe)
  - Office-based Specialist in vascular medecine, Troyes
  - Office-based Specialist in vascular medecine, Valence
  - Office-based Specialist in vascular medecine, Vannes
  - Office-based Specialist in vascular medecine, Vendôme
  - Office-based Specialist in vascular medecine, Verrières-le-Buisson
  - Office-based Specialist in vascular medecine, Versailles
  - Office-based Specialist in vascular medecine, Vesoul
  - Office-based Specialist in vascular medecine, Vénissieux
  - Office-based Specialist in vascular medecine, Vichy
  - Office-based Specialist in vascular medecine, Vienne
  - Office-based Specialist in vascular medecine, Villebon-sur-Yvette
  - Office-based Specialist in vascular medecine, Villefranche-sur-Saône
  - Office-based Specialist in vascular medecine, Villemoisson-sur-Orge
  - Office-based Specialist in vascular medecine, Villeurbanne
  - Office-based Specialist in vascular medecine, Vincennes
  - Office-based Specialist in vascular medecine, Viroflay
  - Office-based Specialist in vascular medecine, Vizille
  - Office-based Specialist in vascular medecine, Voiron
  - Office-based Specialist in vascular medecine, Wissembourg
  - Office-based Specialist in vascular medecine, Wizernes
- Office-based Specialist in vascular medecine, Basse-Terre, Guadeloupe

REFERENCES:
- [Background] Bosson JL, Labarere J, Sevestre MA, Belmin J, Beyssier L, Elias A, Franco A, Le Roux P. Deep vein thrombosis in elderly patients hospitalized in subacute care facilities: a multicenter cross-sectional study of risk factors, prophylaxis, and prevalence. Arch Intern Med. 2003 Nov 24;163(21):2613-8. doi: 10.1001/archinte.163.21.2613. PMID 14638561
- [Background] Samama MM. An epidemiologic study of risk factors for deep vein thrombosis in medical outpatients: the Sirius study. Arch Intern Med. 2000 Dec 11-25;160(22):3415-20. doi: 10.1001/archinte.160.22.3415. PMID 11112234
- [Background] Goldhaber SZ, Visani L, De Rosa M. Acute pulmonary embolism: clinical outcomes in the International Cooperative Pulmonary Embolism Registry (ICOPER). Lancet. 1999 Apr 24;353(9162):1386-9. doi: 10.1016/s0140-6736(98)07534-5. PMID 10227218
- [Background] Stein PD, Hull RD, Ghali WA, Patel KC, Olson RE, Meyers FA, Kalra NK. Tracking the uptake of evidence: two decades of hospital practice trends for diagnosing deep vein thrombosis and pulmonary embolism. Arch Intern Med. 2003 May 26;163(10):1213-9. doi: 10.1001/archinte.163.10.1213. PMID 12767959
- [Background] Sevestre MA, Labarere J, Brin S, Carpentier P, Constans J, Degeilh M, Deslandes B, Elgrishi I, Lanoye P, Laroche JP, Le Roux P, Pichot O, Quere I, Bosson JL; OPTIMEV study. [Optimizing history taking for evaluating the risk of venous thromboembolism: the OPTIMEV study]. J Mal Vasc. 2005 Sep;30(4 Pt 1):217-27. doi: 10.1016/s0398-0499(05)88206-x. French. PMID 16292199
- [Derived] Galanaud JP, Arnoult AC, Sevestre MA, Genty C, Bonaldi M, Guyard A, Giordana P, Pichot O, Colonna M, Quere I, Bosson JL; OPTIMEV-SFMV Investigators. Impact of anatomical location of lower limb venous thrombus on the risk of subsequent cancer. Thromb Haemost. 2014 Dec;112(6):1129-36. doi: 10.1160/TH14-04-0351. Epub 2014 Aug 7. PMID 25104514
- [Derived] Le Moigne E, Genty C, Meunier J, Arnoult AC, Righini M, Bressollette L, Bosson JL, Le Gal G; OPTIMEV Investigators. Validation of the LEFt score, a newly proposed diagnostic tool for deep vein thrombosis in pregnant women. Thromb Res. 2014 Sep;134(3):664-7. doi: 10.1016/j.thromres.2014.07.009. Epub 2014 Jul 17. PMID 25087889
- [Derived] Galanaud JP, Bosson JL, Genty C, Presles E, Cucherat M, Sevestre MA, Quere I, Decousus H, Leizorovicz A. Superficial vein thrombosis and recurrent venous thromboembolism: a pooled analysis of two observational studies. J Thromb Haemost. 2012 Jun;10(6):1004-11. doi: 10.1111/j.1538-7836.2012.04704.x. PMID 22429908
- [Derived] Galanaud JP, Sevestre MA, Genty C, Laroche JP, Zizka V, Quere I, Bosson JL; OPTIMEV SFMV investigators. Comparison of the clinical history of symptomatic isolated muscular calf vein thrombosis versus deep calf vein thrombosis. J Vasc Surg. 2010 Oct;52(4):932-8, 938.e1-2. doi: 10.1016/j.jvs.2010.05.019. Epub 2010 Jul 13. PMID 20630688

RESULTS

PARTICIPANT FLOW:
Groups:
- OPTIMEV: patients with suspected Deep Vein Thrombosis (DVT) or Pulmonary Embolism (PE)
Period: Overall Study
Arm/Group | OPTIMEV
Started | 8256
Completed | 4931 (total recruited for the follow up)
Not Completed | 3325
Not completed — ineligible | 17
Not completed — not living in France | 348
Not completed — refused to participate | 189
Not completed — controls randomised for no follow up | 2770
Not completed — missing information inclusion criteria | 1

BASELINE CHARACTERISTICS:
Arm/Group | OPTIMEV
Number analyzed (Participants) | 8256
Age Continuous [Mean (Standard Deviation); unit: years] | 62 (18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5063
  Male | 3193
Region of Enrollment [Number; unit: participants]
  France | 7908
  Guadeloupe | 321
  Belgium | 27

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Developed a New or Recurrence of Venous Thromboembolism (VTE)
Description: new VTE which can occur during follow up for no VTE patients at inclusion. Or VTE recurrence for VTE patients at inclusion.
Time Frame: at 3 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | OPTIMEV
Number analyzed (Participants) | 4931
percentage of participants | 8.94 [8.14 to 9.83]

2. Secondary Outcome: Percentage of Participants Who Developed Major Bleeding Events
Time Frame: at 3 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | OPTIMEV
Number analyzed (Participants) | 4931
percentage of participants | 3.00 [2.54 to 3.54]

3. Secondary Outcome: Percentage of Participants With Treatment Anticoagulant Prescribed
Time Frame: after inclusion
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | OPTIMEV
Number analyzed (Participants) | 4931
percentage of participants | 52.23 [50.82 to 53.63]

4. Secondary Outcome: Percentage of Participants Who Developed Cardiovascular Events
Time Frame: at 3 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | OPTIMEV
Number analyzed (Participants) | 4931
percentage of participants | 6.98 [6.26 to 7.77]

5. Secondary Outcome: Percentage of Participants Who Died From Any Cause
Time Frame: at 3 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | OPTIMEV
Number analyzed (Participants) | 4931
percentage of participants | 17.0 [15.9 to 18.0]

6. Secondary Outcome: Percentage of Participants Who Developed Cancer Onset
Time Frame: at 3 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | OPTIMEV
Number analyzed (Participants) | 4931
percentage of participants | 4.10 [3.56 to 4.73]

7. Secondary Outcome: Percentage of Participants Who Developed Venous Insufficiency (Leg Ulcer)
Time Frame: at 3 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | OPTIMEV
Number analyzed (Participants) | 4931
percentage of participants | 0.34 [0.20 to 0.55]

ADVERSE EVENTS:
Arm/Group | OPTIMEV
Serious Adverse Events (participants affected / at risk) | 1147/4931
Other Adverse Events (participants affected / at risk) | 273/4931
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | OPTIMEV (N=4931)
death (General disorders) | 822 — Validation by an expert committee
cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 182 — Validation by an expert committee
cardiovascular (Cardiac disorders) | 310 — Validation by an expert committee
haemorrhage (Blood and lymphatic system disorders) | 135 — Validation by an expert committee
Pulmonary Embolism (PE) (Vascular disorders) | 122 — Pulmonary Embolism (PE) with Deep Vein Thrombosis (DVT) or not. Validation by an expert committee
OTHER ADVERSE EVENTS (reported when occurring in more than 0.1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | OPTIMEV (N=4931)
Deep Vein Thrombosis (DVT) (Vascular disorders) | 186 — Validation by an expert committee
Superficial Vein Thrombosis (SVT) (Vascular disorders) | 81 — Validation by an expert committee
Upper Deep Vein Thrombosis (Vascular disorders) | 6 — Validation by an expert committee

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The protocol OPTIMEV will follow the international recommendations: "Uniforms Requirements for Manuscripts Submitted to Biomedical Journals" (http://www.icmje.org)